CLINICAL TRIAL: NCT01329354
Title: Phase II Clinical Trial of Immunotherapy With Rituximab and Autologous Effector Lymphocytes in Patients With Non-Hodgkin Follicular Lymphoma in Response to First Line Chemotherapy
Brief Title: Rituximab and Autologous Effector Lymphocytes in Non-Hodgkin Follicular Lymphoma in Response to First Line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LFNK; 2009-017829-19 (EudraCT Number)
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Follicular Lymphoma; Follicular Non-Hodgkin´s Lymphoma; Autologous Effector Lymphocytes
Keywords: Follicular lymphoma; Follicular non-Hodgkin´s lymphoma; Autologous effector lymphocytes; Cell Therapy; Maintenance therapy; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — CD83 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous effector lymphocytes (Experimental)
  Interventions: Biological: Autologous effector lymphocytes expanded ex-vivo

INTERVENTIONS:
Biological: Autologous effector lymphocytes expanded ex-vivo — Maintenance therapy with Rituximab every two months is the standard of care for patients with follicular lymphoma after induction therapy. The intervention consists on the administration of autologous effector lymphocytes expanded ex-vivo every two Rituximab administrations.
  Other Names: LAK; LAK cells; Activated lymphocytes

SUMMARY:
Nowadays, therapy with monoclonal antibodies is considered to be a standard treatment that increases the rate of remissions and the overall survival in patients with follicular lymphoma. Nevertheless there are an important number of patients who do not benefit from this therapy. A way to improve the efficiency of monoclonal antibodies therapy could be to improve the activity of the effector arm of the immune system. A strategy that has been proposed to obtain this improvement is the utilization of lymphocyte activated killer (LAK) cells. In addition, the combination of LAK cells with monoclonal antibodies might obtain an additive effect across the stimulation of the antibody dependent cellular cytotoxicity (ADCC)activity.

The present clinical assay proposes to study the feasibility, safety and effectiveness of treatment with autologous effector cells expanded ex vivo associated with a standard maintenance treatment with rituximab in patients with follicular lymphoma in remission after first-line treatment. In addition, we plan to analyse various biological parameters that can predict the susceptibility of patients to treatment with rituximab. Specifically, we propose to study the polymorphisms of Fc receptor, polymorphisms related to the ability of complement activation, to study both the complement activity and peripheral blood cell subpopulations that can mediate directly or indirectly dependent antibody cytotoxic effect. We will also try to correlate any of these biological parameters with the response to treatment.

DETAILED DESCRIPTION:
There are many mechanisms involved in the antitumor effect of the antibodies including the induction of apoptosis, blocking angiogenesis, blockade of intracellular signaling pathways, and activation of complement leading to lysis of tumor cells. However it appears that the antibody-dependent cellular cytotoxicity (ADCC) is one of the predominant mechanisms of action. It is important to note that in order to obtain a powerful ADCC effect it is necessary the action of the antibody but also the activity of the effector cell, and thus the competence of the immune system of the guest. There are different cellular subpopulations that mediate the ADCC effect. CTL and NK are two of these subpopulations that can be reduced in patients with cancer.

A way to improve the efficiency of the monoclonal antibodies would be to improve the activity of the effector arm of the immune system. A strategy that that has been planed is the utilization of LAK cells. The culture of lymphocytes of peripheral blood with IL-2 activates the subpopulations of killer cells. This population of killer cells activated with cytokines (LAK: lymphokine activated killer) has a high number of NK and CTL cells, both with increased cytotoxic capacity. It has been demonstrated that the immunotherapy with LAK cells might be an effective and sure treatment for patients with follicular lymphoma.

In a murine model it has been demonstrated that LAK cells associated with monoclonal antibodies increase the antitumoral activity when compared to the administration of antibodies alone. In addition, in this model the combination was also superior to the administration of monoclonal antibodies + IL-2 (Schultz et al., 1990). Other investigators have demonstrated similar results. This information supports the idea of the combined therapy consisting in LAK with anti-CD20 antibodies. This therapy can induce a destruction of CD20 positive cells greater than that with the monoclonal antibodies alone. In addition, it has been reported that the administration of systemic IL-2 and LAK cells improves the ADCC in lymphoma patients treated with rituximab. It is a small pilot study, with 10 patients. Seven of them received LAK cells following a programmed way. The safety of the treatment and the promising results demonstrated in this study encourage to investigate in this line.

Since one of the mechanisms of action of the monoclonal antibodies is to promote ADCC , our hypothesis is that the treatment with a suspension of autologous effector lymphocytes expanded ex-vivo with culture should modify the biological effect of the treatment with rituximab in follicular lymphoma patients, with an acceptable safety profile, and probably increasing the efficiency of the monoclonal antibodies. In order to evaluate this hypotesis we propose an open, prospective, historically controlled, phase II clinical study in patients with follicular lymphoma who have achieved a remission after first-line therapy including the anti-CD20 monoclonal antibody rituximab and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed follicular lymphoma CD20-positive grade 1, 2 ó 3a.
* Patients with aptitude to sign the written informed consent and to express his desire to fulfill all the requirements of the protocol during the period of study.
* Patients not treated before. The induction treatment with rituximab and chemotherapy must be the first line for the patients who are included in the study.
* Patients undergoing maintenance therapy with rituximab every two/three months.
* Ann Arbor stage II, III o IV before receiving the induction treatment with rituximab and chemotherapy.
* The patient must have achieved a partial or complete response based on the revised International Workshop Response Criteria (IWRC) (Cheson, et al 2007) following the induction treatment.
* Age >18 years and <75 years.
* Performance status <2 following the Eastern Cooperative Oncology Group (ECOG).
* Screening laboratory values obtained 28 days before registry (unless due to lymphoma involvement of the bone marrow): Hemoglobin > 8,0 g/dL (5,0 mmol/L), Neutrophil absolute count > 1,5 x 109/L,Platelets > 100 x 109/L

Exclusion Criteria:

* Patients with transformed follicular lymphoma into diffuse large B-cell lymphoma.
* Patients with evidence of follicular lymphoma grade 3b.
* Patients with evidence of primary cutaneous or gastrointestinal follicular lymphoma.
* Patients with evidence of current central nervous system involvement.
* Patients who received previous induction treatment other than rituximab and chemotherapy.
* Patients receiving chronic immunosuppressive agents in the last 4 weeks. Patients may be receiving stable chronic doses of corticosteroids with a maximum dose of 20 mg/day of prednisone or equivalent.
* Patients who have a history of another primary malignancy < 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix.
* Decompensated renal function: serum creatininea > 2,0 mg/dL (197 u.mol/L.
* Decompensated hepatic function: total bilirrubine > 2,0 mg/dL (34 umol/L), AST (SGOT) > 3 x ULN, unless due to lymphoma involvement
* Patients with a known history of human immunodeficiency virus (HIV) seropositivity, chronic hepatitis or other active viral infections due to hepatitis B virus (HBV) or hepatitis C virus (HVC).
* Patients with underlying serious diseases that in the criteria of the investigator could concern the capacity of the patient to take part in the test (for example, infection in process, not controlled diabetes mellitus, gastric ulcers, autoimmune active disease).
* Life expectancy <6 months.
* Female patients who are pregnant or breast feeding.
* Patients with known hypersensitivity to rituximab or other murine proteins or to any of the excipients.
* Patients who are using other investigational agents or who have received investigational drus 30 days prior to study drug start.
* Any other medical or psychological coexistent condition that rejects the participation in the study or compromises the aptitude to give the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2011-03; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) from the entry in the study. | 01/03/2015
  The PFS is defined as the time from the entry in the study up to the progression of the disease.

SECONDARY OUTCOMES:
Event free survival from the entry in the study | 01/03/2015
  Event: progression, relapse, death for any reason, or institution of a new anti-lymphoma treatment (chemotherapy, radiotherapy or immunotherapy).
Time to the next anti-lymphoma treatment | 01/03/2015
  Defined as the time from the registry of the patient up to the institution of a new regimen (chemotherapy, radiotherapy or immunotherapy).
Disease free survival | 01/03/2015
  Defined as the time from the first complete response documented up to the relapse
Safety | 01/01/2012
  Defined as the incidence of toxicity of all the treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Panizo, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Garcia-Munoz R, Lopez-Diaz-de-Cerio A, Feliu J, Panizo A, Giraldo P, Rodriguez-Calvillo M, Grande C, Pena E, Olave M, Panizo C, Inoges S. Follicular lymphoma: in vitro effects of combining lymphokine-activated killer (LAK) cell-induced cytotoxicity and rituximab- and obinutuzumab-dependent cellular cytotoxicity (ADCC) activity. Immunol Res. 2016 Apr;64(2):548-57. doi: 10.1007/s12026-015-8747-9. PMID 26659089